CLINICAL TRIAL: NCT06465121
Title: Difficult Venous Access in Pediatric Patients: Paramedical Care Using Ultrasound Guidance
Brief Title: Difficult Intravenous Access in Pediatric Patients: Paramedical Care Using Ultrasound Guidance
Acronym: VVParamECHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PP24044*
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Catheter Related Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guidance (Experimental): peripheral intravenous catheterization performed with ultrasound guidance by a trained nurse
  Interventions: Procedure: peripheral intravenous catheterization performed with ultrasound guidance by a trained nurse
- Standard of care (No Intervention): Peripheral intravenous catheterization by visualization and palpation of the vein alone

INTERVENTIONS:
Procedure: peripheral intravenous catheterization performed with ultrasound guidance by a trained nurse — Intravenous catheterization using ultrasound-guidance to allow real-time visualization of target veins in pediatric patients with difficult intravenous access
  Arms: Ultrasound guidance

SUMMARY:
Obtaining intravenous access is difficult in the pediatric population. Ultrasound-guidance allows real-time visualization of target veins which are invisible and impalpable. We hypothesize that the use of ultrasound by a trained nurse team would improve the success rate of peripheral intravenous catheter insertion in pediatric patients with difficult intravenous access, compared to palpation of the vein alone.

For this study, when peripheral intravenous catheterization will be indicated in one of the participating pediatric services for an eligible patient, state-certified nurse investigators, trained in ultrasound guidance, will be contacted. After verification of eligibility criteria and all informed consents obtained, one of the investigators will randomize the patient in one of the 2 treatment groups under study: peripheral intravenous catheterization by visualization and palpation of the vein alone (standard of care) or by ultrasound guidance performed by a trained nurse.

Several outcomes will be measured and compared between the 2 groups (e.g. successful insertion of intravenous catheter, pain, adverse events).

DETAILED DESCRIPTION:
Venipunctures are very common in hospitalized patients. Obtaining venous access is more difficult in the pediatric population, particularly due to the smaller size of the vessels and the more difficult cooperation of patients. Traditional method for inserting intravenous catheter access requires knowledge of vascular anatomy to estimate the location of the target vein and requires visualization or palpation of the vein. The success rate for peripheral intravenous catheterization in pediatric patients is approximately 60% after one attempt and 90% after four. Delays in intravenous access can result in significant morbidity and mortality. Thus, alternative methods should be considered to improve pediatric access sites.

Ultrasound-guidance allows real-time visualization of target veins which are invisible and impalpable. We hypothesize that the use of ultrasound by a trained nurse team would improve the success rate of peripheral intravenous catheter insertion in pediatric patients with difficult intravenous access. This could also have an impact on the frequency of the main associated adverse events.

For this study, when peripheral intravenous catheterization will be indicated in one of the participating pediatric services for an eligible patient, state-certified nurse investigators, trained in ultrasound guidance, will be contacted. After verification of eligibility criteria and all informed consents obtained, one of the investigators will randomize the patient in one of the 2 treatment groups under study: peripheral intravenous catheterization by visualization and palpation of the vein alone (standard of care) or by ultrasound guidance performed by a trained nurse.

Several outcomes will be measured and compared between the 2 groups (e.g. successful insertion of intravenous catheter, pain, adverse events).

Children will be followed for a maximum of 7 days or until discharge from hospitalization.

ELIGIBILITY:
Inclusion Criteria :

* age ≥ 1 month and < 18 years
* intravenous catheter insertion indicated for hospital care
* DIVA (Difficult Intravenous Access Scale) score ≥ 4
* hospitalized in one of the pediatric departments of the Reims University Hospital
* who agree to participate in the study (if old enough to understand) and for whom the consent of the holder(s) of parental authority has been obtained
* affiliated to a social security scheme

Exclusion Criteria:

* Newborns (< 1 month) and premature babies hospitalized in neonatal intensive care, neonatology and maternity units
* Known vascular pathology
* Hemodialysis with arteriovenous fistula
* Unstable hemodynamic and/or respiratory clinical state according to the judgment of the medical team

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with success at first intravenous catheter insertion attempt | Day 0
  Success at first attempt of intravenous catheter insertion with ultrasound-guidance compared to standard of care for pediatric patients with difficult venous access

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided